CLINICAL TRIAL: NCT00912912
Title: Phase II Study of Sunitinib Malate in Refractory Germ Cell Tumors
Brief Title: Sunitinib Malate in Refractory Germ Cell Tumors
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0685; NCI-2012-01645 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2009-06-01; First posted 2009-06-03 (Estimated); Results first posted 2016-01-27 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-03

CONDITIONS: Genitourinary Disease
Keywords: Genitourinary; Testis; Refractory Germ Cell Tumors; Advanced germ cell tumors; GCTs; Sunitinib Malate; Sutent; SU011248
MeSH Terms: conditions — Urogenital Diseases; Neoplasms, Germ Cell and Embryonal | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sunitinib Malate (Experimental): Sunitinib Malate 50 mg capsules once a day (by mouth) for 4 weeks in a row in a 6 week cycle.
  Interventions: Drug: Sunitinib Malate

INTERVENTIONS:
Drug: Sunitinib Malate — 50 mg capsules once a day (by mouth) for 4 weeks in a row in a 6 week cycle.
  Other Names: SU011248; Sutent

SUMMARY:
The goal of this clinical research study is to learn if Sutent® (sunitinib malate, SU011248) can control the disease in patients with germ cell tumors that are resistant to earlier treatment.

DETAILED DESCRIPTION:
The Study Drug:

Sunitinib malate is designed to block pathways that control important events such as the growth of blood vessels that are essential for the growth of cancer.

Within 14 days of enrollment on this study, you will have the following tests and procedures performed:

* Your complete medical history will be recorded.
* You will have a physical exam.

Within 7 days of enrollment on this study, you will have the following tests and procedures performed:

-Blood (about 3 teaspoons) and urine will be collected for routine testing and to test for certain biomarkers (to check the status of the disease).

Study Drug Administration:

If you are found to be eligible to take part in this study, you will take sunitinib malate capsules once a day (by mouth) for 4 weeks in a row followed by 2 weeks with no study drug. These 6 weeks are considered 1 cycle of study treatment.

Study Visits:

On Day 1 of each cycle (about every 6 weeks), you will have the following tests done before you take the study drug:

* You will have a physical exam.
* You will be asked about how you are feeling and about any side effects you have experienced since your last visit.
* You will have blood (about 3 teaspoons) and urine collected for routine tests and to test for certain biomarkers.

For the first 4 weeks of treatment, you should have your blood pressure monitored. This may be done at your home with a digital pressure device, or you may visit your local doctor for this testing.

About Day 21 of Cycles 1 and 2, blood (about 2- 3 teaspoons) will be drawn for routine tests. This may be done at your local doctor's office and results faxed to the study doctor.

On Day 1 of Cycle 2, Day 1 of Cycle 3, and then Day 1 of every 2 cycles after that (Cycle 5, Cycle 7, and so on), you will have imaging scans to check status of the disease. This could include CT or MRI scans, an ECG, and a chest x-ray. If your doctor thinks it is necessary, you may have additional imaging scans at any time.

On Day 1 of every other cycle (Cycle 3, Cycle 5, and so on), you will have an echocardiogram or MUGA scan.

Length of Study:

You may remain on study for as long as you are benefitting. You will be taken off study if intolerable side effects occur or if the disease gets worse. However, if the disease gets worse very quickly during Cycles 1 or 2, you will be taken off study at that time.

Off-Study Visit:

When you are taken off of treatment on this study, the following tests and procedures will be performed:

* You will have a physical exam.
* You will be asked how you are feeling and about any changes in your medical history since beginning this study.
* You will also be asked about any side effects you have experienced since your last visit.

This is an investigational study. Sunitinib malate is approved by the FDA for the treatment of adults with kidney cancer. Its use in patients with germ cell tumors is investigational. Up to 42 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Progressive metastatic Germ-cell tumors (GCTs) of gonadal or extragonadal origin in males after failure of front-line therapy and at least one salvage regimen.
2. Must have evaluable or measurable disease by clinical or radiological studies. Alternatively, in the absence of radiologically evaluable or measurable disease, two sequentially rising marker values each one week apart attributed by treating physician to germ cell tumor is permitted; either beta human chorionic gonadotropin (hCG) above 50 mIU/ml and/or alpha-fetoprotein (AFP) above 20 ng/ml qualifies as eligible.
3. The Eastern Cooperative Oncology Group (ECOG) Performance Score 0-2
4. Adequate organ function as follows: Calculated creatinine clearance >/= 35cc/min, Absolute neutrophil count >/= 1500/mm^3, hemoglobin >/= 8 g/dL, serum calcium </= 12 mg/dL, Platelet count >/= 75,000/mm^3, AST (SGOT)/ALT (SGPT) < 2.5 x upper limit of normal (ULN), Total bilirubin < 2.0mg/dl.
5. Resolution of all acute toxic effects of prior chemotherapy or radiotherapy or surgical procedures to NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0 grade </= 2.
6. At least 18 years of age as safety of sunitinib in a pediatric population has not been established.
7. Able to provide informed consent
8. Must be able to ingest oral medication
9. Male subjects must be surgically sterile or must agree to use effective contraception during the period of therapy. The definition of effective contraception will be based on the judgment of the principal investigator or a designated associate.
10. Patients who have not received prior high-dose chemotherapy and stem cell rescue as salvage therapy will have this option discussed with them. Only patients ineligible, unwilling or unable to undertake this option will be eligible for this trial.

Exclusion Criteria:

1. NCI CTCAE Version 3.0 grade 3 hemorrhage within the 4 weeks prior to starting the study treatment.
2. Any of the following within the 12 months prior to study drug administration: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack, or pulmonary embolism.
3. Patients with history of Long QT syndrome.
4. Ongoing cardiac dysrhythmias of NCI CTCAE Version 3.0 grade >/= 2.
5. Uncontrolled Hypertension (> 140/90 mm Hg despite optimal medical therapy).
6. Pre-existing thyroid abnormality with thyroid function that cannot be maintained in the normal range with medication.
7. Symptomatic bowel obstruction.
8. Prior VEGFR/PDGFR inhibitor therapy.
9. Known human immunodeficiency virus infection, chronic active hepatitis or liver cirrhosis.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2009-05; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lance Pagliaro, MD, BA, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Subbiah V, Meric-Bernstam F, Mills GB, Shaw KR, Bailey AM, Rao P, Ward JF, Pagliaro LC. Next generation sequencing analysis of platinum refractory advanced germ cell tumor sensitive to Sunitinib (Sutent(R)) a VEGFR2/PDGFRbeta/c-kit/ FLT3/RET/CSF1R inhibitor in a phase II trial. J Hematol Oncol. 2014 Aug 1;7:52. doi: 10.1186/s13045-014-0052-x. PMID 25085632
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: May 29, 2009 to July 29, 2010. All recruitment was done at The University of Texas (UT) MD Anderson Cancer Center.
Pre-assignment Details: Study was closed early due to low rate of response and slow accrual.
Period: Overall Study
Arm/Group | Sunitinib Malate
Started | 5
Completed | 1
Not Completed | 4
Not completed — Withdrawal by Subject | 1
Not completed — Disease Progression | 3

BASELINE CHARACTERISTICS:
Arm/Group | Sunitinib Malate
Number analyzed (Participants) | 5
Age, Continuous [Median (Full Range); unit: years] | 29 [17 to 36]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: 12 Week Progression Free Survival Rate in Refractory Germ Cell Tumors Treated With Sunitinib Malate
Description: Measurable disease or response recorded from start of treatment until disease progression/recurrence. Participants who die during therapy or are lost to follow-up shall be counted as progressive disease. Progressive disease defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since the treatment started or the appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions. Evaluation of measurable disease response follows Response Evaluation Criteria in Solid Tumors (RECIST) guidelines.
Time Frame: 12 weeks
Measure: Number; unit: Percentage of Participants
Arm/Group | Sunitinib Malate
Number analyzed (Participants) | 5
Percentage of Participants | 20

ADVERSE EVENTS:
Time Frame: Adverse event collection through each cycle, defined as a planned 6-week treatment interval (cycle) with participants to complete at least 2 cycles of therapy unless evidence of rapid disease progression.
Arm/Group | Sunitinib Malate
Serious Adverse Events (participants affected / at risk) | 3/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sunitinib Malate (N=5)
PAIN (MID-BACK) (Musculoskeletal and connective tissue disorders) | 1 (1)
PAIN (LEFT-CHEST) (General disorders) | 1 (1)
PAIN (THORACIC BACK) (Musculoskeletal and connective tissue disorders) | 1 (1)
HEADACHE (Nervous system disorders) | 1 (1)
HEMORRHAGE (Vascular disorders) | 1 (1)
DEATH (General disorders) | 1 (1)
WEAKNESS (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sunitinib Malate (N=5)
CONSTIPATION (Gastrointestinal disorders) | 2 (7)
MOOD ALTERATION (DEPRESSION) (Psychiatric disorders) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 3 (5)
VOMITING (Gastrointestinal disorders) | 2 (7)
FATIGUE (General disorders) | 4 (17)
NEUROPATHY: SENSORY (Nervous system disorders) | 4 (5)
INSOMNIA (General disorders) | 1 (1)
PAIN (OTHER) (General disorders) | 2 (3)
PAIN (EXTREMITY - LIMB) (Musculoskeletal and connective tissue disorders) | 2 (2)
PAIN (ABDOMEN) (Gastrointestinal disorders) | 3 (4)
ALOPECIA (Skin and subcutaneous tissue disorders) | 2 (2)
HEMOGLOBIN (Blood and lymphatic system disorders) | 4 (9)
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1)
ANOREXIA (Gastrointestinal disorders) | 2 (5)
RASH/DESQUAMATION (Skin and subcutaneous tissue disorders) | 3 (4)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 2 (4)
DIARRHEA (Gastrointestinal disorders) | 2 (3)
HYPOPIGMENTATION (Skin and subcutaneous tissue disorders) | 2 (4)
WEIGHT LOSS (General disorders) | 1 (1)
PAIN (CHEST/THORAX) (General disorders) | 2 (2)
SUPRAVENTRICULAR AND NODAL ARRHYTHMIA (Cardiac disorders) | 2 (2)
PLATELETS (Blood and lymphatic system disorders) | 3 (4)
NEUTROPHILS/GRANULOCYTES (Blood and lymphatic system disorders) | 3 (3)
BRUISING (Skin and subcutaneous tissue disorders) | 1 (1)
PAIN (BACK) (Musculoskeletal and connective tissue disorders) | 2 (2)
HYPOMAGNESEMIA (Metabolism and nutrition disorders) | 2 (2)
PROTEINURIA (Metabolism and nutrition disorders) | 2 (2)
HEADACHE (Nervous system disorders) | 1 (1)
ULCER - GI (Gastrointestinal disorders) | 1 (1)
CREATININE (Metabolism and nutrition disorders) | 1 (1)
HYPERBILIRUBINEMIA (Metabolism and nutrition disorders) | 1 (5)
LYMPHOPENIA (Blood and lymphatic system disorders) | 1 (2)
HYPOTHYROIDISM (Endocrine disorders) | 1 (1)
MUSCULOSKELETAL/SOFT TISSUE - OTHER (Musculoskeletal and connective tissue disorders) | 1 (1)
DRY SKIN (Skin and subcutaneous tissue disorders) | 1 (2)
GASTROINTESTINAL - OTHER (Gastrointestinal disorders) | 1 (1)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 1 (1)
ENDOCRINE - OTHER (Endocrine disorders) | 1 (1)
NEUROLOGY - OTHER (Nervous system disorders) | 1 (2)
MUCOSITIS/STOMATITIS (Gastrointestinal disorders) | 4 (13)
LEUKOCYTES (Blood and lymphatic system disorders) | 4 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes